CLINICAL TRIAL: NCT03919734
Title: Morbidity and Mortality in Patients With Adrenal Incidentalomas With and Without Autonomous Cortisol Secretion
Brief Title: Morbidity and Mortality in Autonomous Cortisol Secretion
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Henrik Olsen, Principal Investigator Henrik Olsen, MD, PhD., Region Skane
Other Study IDs: 1
Record Dates: First submitted 2019-04-07; First posted 2019-04-18 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Adrenal Incidentaloma; Cortisol Overproduction
MeSH Terms: conditions — Adrenal incidentaloma; ACTH Syndrome, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- AI ACS/possible ACS: Patients with adrenal incidentalomas and cortisol following overnight 1-mg dexamethasone suppression equal to or above 50 nmol/l. The patients should not have clinical signs of Cushing Syndrome, such as catabolic skin and muscle changes.
- AI non-ACS: Patients with adrenal incidentalomas and cortisol following overnight 1-mg dexamethasone suppression below 50 nmol/l.
- Treatment with Inhalation Steroids: Patients treated with inhalation steroids with and without ACS/possible ACS but not operated with adrenalectomy.
- Adrenalectomy: Patients with unilateral AI operated with adrenalectomy
- Controls: A Group of Controls matched for sex and age, achieved by the government agency "Statistics Sweden" (SCB).

SUMMARY:
Benign enlargements of the adrenal glands (adrenal adenomas) are frequent in adults. In the general population these adenomas are rare in subjects below 40 years of age but at the age of 60 and 80 years the prevalence is 6 and 8-10 % respectively. Since these adenomas do not causes obvious symptoms they are almost exclusively found incidentally in patients examined radiologically for other reasons than suspected adrenal disease. These enlargements are thus termed adrenal incidentalomas (AI). AI may secrete cortisol and more than 25 percent of patients with an AI have increased cortisol levels called autonomous cortisol secretion (ACS). Such increased secretion of cortisol may cause metabolic complications such as hypertension, high cholesterol, diabetes and cardiovascular disease. Studies have shown that ACS may cause increased mortality. These studies are however small and have not adequately taking other conditions into account which most likely influences the result.

The investigators hypothesis is that ACS is linked to increased mortality as the previous studies have shown. The aim is to perform a larger study on patients with adrenal incidentalomas, both with and without ACS, and compare the mortality rates with a control group matched for age and sex. This study may more precisely describe the cardiovascular risk for ACS and define the risk at different levels of ACS.

DETAILED DESCRIPTION:
Patients with adrenal adenomas may have autonomous cortisol secretion (ACS) that has been linked to hypertension, diabetes, dyslipidemia and cardiovascular disease. Patients with ACS also have been found to have increased mortality. In two studies the excess mortality was caused by cardiovascular disease and in one study by cancer.

ACS is diagnosed by increased cortisol (≥50 nmol/l) following 1-mg dexamethasone suppression (DST) often in combination with another confirmatory test such as low ACTH, increased urinary cortisol, increased midnight salivary cortisol or a dexamethasone suppression test with a higher dexamethasone dose. Cortisol secretion from an AI has been considered exclusively autonomous but the investigators have recently shown that a large group of patients with normal results on DST have low ACTH indicating that another factor than ACS may suppress the HPA-axis. The hypothesis is that these patients have an increased sensitivity to ACTH, which results in lower ACTH levels. It has however not been studied whether the increased sensitivity to ACTH is linked to increased cardiovascular morbidity and mortality.

Patient data is collected from the patient cards and radiology images. Patients are included according to the eligibility criteria. The patients will be separated in the following groups:

1. No ACS, inhalation steroids or adrenalectomy.
2. ACS/possible-ACS but not treatment with inhalation steroids or adrenalectomy
3. Treatment inhalation steroids but not operated.
4. Unilateral AI and treated with adrenalectomy but no inhalation steroids. The group is separated in patients without ACS and patients with possible ACS/ACS.

Three age and gender matched subjects from the general population for every patient will serve as a controls.

Outcome data on patients and controls is received from The National Board of Health and Welfare. The control group is achieved from SCB, Sweden (Statistics Sweden). The following outcome data will be collected: Data on mortality, cause of mortality and inpatient and outpatient cardiovascular diagnoses. The study design reduces the risk for bias between the clinical endpoints and the patient's cortisol and ACTH levels. The patient cohorts will be finally defined before the investigators receive the clinical endpoints from The National Board of Health and Welfare.

Statistical analysis: The prevalence of the outcome data in the groups of patients will be compared. The investigators will adjusted for differences between the groups in sex, age, smoking, impaired renal function, and existing cardiovascular disease.

The following variables will be examined in relation to the outcome data: Cortisol following dexamethasone (≥50 nmol/l, ≥83 nmol/l and ≥138 nmol/l), low basal ACTH (<2.0 pmol/l), DHEAS, the size of the AI and bilateral versus unilateral AI.

Study Status: We anticipate to receive the outcome data from The National Board of Health and Welfare in October 2019. The study has thus been slightly delayed. Data on morbidity will only be available until December 31, 2017 due to a delay in reporting to The National Board of Health and Welfare. The secondary outcome measure has been changed to a composite of cardiovascular endpoints.

ELIGIBILITY:
Inclusion Criteria:

Patients with adrenal incidentalomas examined at Skane University Hospital and Helsingborg Hospital during the period from January 1, 2005 to September 15, 2015.

Exclusion Criteria:

1. Size of incidentaloma below 1 cm
2. Malignant disease with metastases,
3. Incidentaloma not an adenoma but for example malignancy, myelolipoma and bleedings
4. Pheochromocytomas
5. Primary aldosteronism
6. Continuous treatment with systemic glucocorticoid under the last 3 months.
7. Cushing Syndrome
8. Medication affecting dexamethasone metabolism.
9. Treatment with systemic estrogen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients examined at the Endocrine outpatient ambulatory first time for adrenal incidentalomas during the period from January 1, 2005 to September 15, 2015.
  A Group of Age and sex matched controls developed by SCB.
Sampling Method: Non-Probability Sample
Enrollment: 4596 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Number of patients deceased, both totally and divided into three specified diagnose groups (cardiovascular disease, infections and cancer). | From date of enrollment until December 31, 2018.
  The cause of death is defined by the ICD-10 code reported by The National Board of Health and Welfare.

SECONDARY OUTCOMES:
A composite of cardiovascular death, nonfatal myocardial infarction (excluding silent myocardial infarction), nonfatal stroke, hospitalization for heart failure and revascularization (CABG and PCI). The endpoints will also be calculated separately. | From date of enrollment until December 31, 2017.
  The diagnoses is defined by the ICD-10 code and Swedish classification of healthcare interventions (KVÅ-codes FNA-FNG) both reported by The National Board of Health and Welfare

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Olsen, MD, PhD, Principal Investigator — Medical Faculty, University of Lund
Locations (1):
- Dept. of Endocrinology, Skåne University Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fassnacht M, Arlt W, Bancos I, Dralle H, Newell-Price J, Sahdev A, Tabarin A, Terzolo M, Tsagarakis S, Dekkers OM. Management of adrenal incidentalomas: European Society of Endocrinology Clinical Practice Guideline in collaboration with the European Network for the Study of Adrenal Tumors. Eur J Endocrinol. 2016 Aug;175(2):G1-G34. doi: 10.1530/EJE-16-0467. PMID 27390021
- [Background] Debono M, Bradburn M, Bull M, Harrison B, Ross RJ, Newell-Price J. Cortisol as a marker for increased mortality in patients with incidental adrenocortical adenomas. J Clin Endocrinol Metab. 2014 Dec;99(12):4462-70. doi: 10.1210/jc.2014-3007. PMID 25238207
- [Background] Di Dalmazi G, Vicennati V, Garelli S, Casadio E, Rinaldi E, Giampalma E, Mosconi C, Golfieri R, Paccapelo A, Pagotto U, Pasquali R. Cardiovascular events and mortality in patients with adrenal incidentalomas that are either non-secreting or associated with intermediate phenotype or subclinical Cushing's syndrome: a 15-year retrospective study. Lancet Diabetes Endocrinol. 2014 May;2(5):396-405. doi: 10.1016/S2213-8587(13)70211-0. Epub 2014 Jan 29. PMID 24795253
- [Background] Patrova J, Kjellman M, Wahrenberg H, Falhammar H. Increased mortality in patients with adrenal incidentalomas and autonomous cortisol secretion: a 13-year retrospective study from one center. Endocrine. 2017 Nov;58(2):267-275. doi: 10.1007/s12020-017-1400-8. Epub 2017 Sep 8. PMID 28887710
- [Background] Olsen H, Kjellbom A, Londahl M, Lindgren O. Suppressed ACTH Is Frequently Unrelated to Autonomous Cortisol Secretion in Patients With Adrenal Incidentalomas. J Clin Endocrinol Metab. 2019 Feb 1;104(2):506-512. doi: 10.1210/jc.2018-01029. PMID 30265354
- [Derived] Kjellbom A, Lindgren O, Danielsson M, Olsen H, Londahl M. Mortality Not Increased in Patients With Nonfunctional Adrenal Adenomas: A Matched Cohort Study. J Clin Endocrinol Metab. 2023 Jul 14;108(8):e536-e541. doi: 10.1210/clinem/dgad074. PMID 36800277
- [Derived] Kjellbom A, Lindgren O, Puvaneswaralingam S, Londahl M, Olsen H. Association Between Mortality and Levels of Autonomous Cortisol Secretion by Adrenal Incidentalomas : A Cohort Study. Ann Intern Med. 2021 Aug;174(8):1041-1049. doi: 10.7326/M20-7946. Epub 2021 May 25. PMID 34029490